CLINICAL TRIAL: NCT04091178
Title: A PHASE II Multicentric Trial Evaluating a High Dose Vitamin D Supplementation to Correct the Vitamin D Deficiency for Breast Cancer Treated by Adjuvant Chemotherapy
Brief Title: Vitamin D Supplementation to Correct the Vitamin D Deficiency for Breast Cancer
Acronym: OPTIVIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICM2013/06
Record Dates: First submitted 2019-09-04; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: A phase 2 clinical trial not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VITAMIN D SUPPLEMENTATION ARM (Experimental): On day 1 of every chemotherapy cycle, the patient will be receive an oral solution of vitamin D (UVEDOSE/calciferol).
  In parallel,a calcium supplementation is prescribed.
  Interventions: Dietary Supplement: VITAMIN D

INTERVENTIONS:
Dietary Supplement: VITAMIN D — ORAL SOLUTION (2 ml) at 100.000 UI

SUMMARY:
An open clinical trial not randomized, multicentric. This study search to evaluate vitamin D supplementation efficacy at high dose (UVEDOSE, colecalciferol, oral solution at 100 000 UI) of vitamin D on day 1 of each cycles for breast cancer treated adjuvant chemotherapy.

A calcium supplementation will be prescribed in parallel.

An initial dosage of 25OH vitamin D rate will be done and a vitamin-calcic dosage will done on day 1 of every cycles of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Breast adenocarcinoma should receive 6 cycles of adjuvant chemotherapy
* Women ≥ 18 years old (no age limit)
* Performance status :0 or 1
* Patients must be affiliated to a Social Security System
* Signed informed consent obtained before any study specific procedures.
* Vitamin D deficiency confirmed ( vitamin D result must be < at 30 ng/ml)

Exclusion Criteria:

* Metastatic disease
* Patients with previous or concomitant other (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years
* calcium or colecalciferol contraindications (vitamin D hypersensitivity - disease or an other condition result in hypercalcaemia or hypercalciuria -Calcic lithiasis- high vitamin D level)
* Presence of the following diseases in the last 3 years : endocrinal disease, A phosphor calcic disorder treated by vitamin D supplementation at 1000 UI/day or more (this patient who have received a dose < 1000 UI/day, will be included after have to stop Vitamin D at least 48 hours ) - Osteopenia or osteoporosis confirmed treated
* Concomittant treatment with an other experimental product
* Pregnant or breastfeeding women
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Normalisation of Vitamin D level | from the Cycle 1 to cycle 6 (each cycle is 21 days)
  percentage of vitamin D level normalisation

SECONDARY OUTCOMES:
initial vitamin D and calcium level | at cycle 1( one cycle is 21 days)
  blood test
normalization of 25-OHD (vitamin D) | at FU 6,12,18,24 months after the first dose of vitamin D
  blood test
adverses events rates | from cycle 1 to follow-up 24 months (one cycle is 21 days)
  graded based on NCI-CTCAE v4.03
vitamin D and calcium level | from cycle 1 to 24 months (one cycle is 21 days)
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: WILLIAM JACOT, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cavalier E, Delanaye P, Chapelle JP, Souberbielle JC. Vitamin D: current status and perspectives. Clin Chem Lab Med. 2009;47(2):120-7. doi: 10.1515/CCLM.2009.036. PMID 19099529
- [Result] Sinotte M, Diorio C, Berube S, Pollak M, Brisson J. Genetic polymorphisms of the vitamin D binding protein and plasma concentrations of 25-hydroxyvitamin D in premenopausal women. Am J Clin Nutr. 2009 Feb;89(2):634-40. doi: 10.3945/ajcn.2008.26445. Epub 2008 Dec 30. PMID 19116321
- [Result] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Result] Bischoff-Ferrari HA, Willett WC, Wong JB, Giovannucci E, Dietrich T, Dawson-Hughes B. Fracture prevention with vitamin D supplementation: a meta-analysis of randomized controlled trials. JAMA. 2005 May 11;293(18):2257-64. doi: 10.1001/jama.293.18.2257. PMID 15886381
- [Result] Tang BM, Eslick GD, Nowson C, Smith C, Bensoussan A. Use of calcium or calcium in combination with vitamin D supplementation to prevent fractures and bone loss in people aged 50 years and older: a meta-analysis. Lancet. 2007 Aug 25;370(9588):657-66. doi: 10.1016/S0140-6736(07)61342-7. PMID 17720017
- [Result] Roux C, Bischoff-Ferrari HA, Papapoulos SE, de Papp AE, West JA, Bouillon R. New insights into the role of vitamin D and calcium in osteoporosis management: an expert roundtable discussion. Curr Med Res Opin. 2008 May;24(5):1363-70. doi: 10.1185/030079908x301857. Epub 2008 Apr 2. PMID 18387220
- [Result] Bischoff-Ferrari HA, Dawson-Hughes B, Willett WC, Staehelin HB, Bazemore MG, Zee RY, Wong JB. Effect of Vitamin D on falls: a meta-analysis. JAMA. 2004 Apr 28;291(16):1999-2006. doi: 10.1001/jama.291.16.1999. PMID 15113819
- [Result] Abbas S, Nieters A, Linseisen J, Slanger T, Kropp S, Mutschelknauss EJ, Flesch-Janys D, Chang-Claude J. Vitamin D receptor gene polymorphisms and haplotypes and postmenopausal breast cancer risk. Breast Cancer Res. 2008;10(2):R31. doi: 10.1186/bcr1994. Epub 2008 Apr 17. PMID 18419802
- [Result] Abbas S, Linseisen J, Slanger T, Kropp S, Mutschelknauss EJ, Flesch-Janys D, Chang-Claude J. Serum 25-hydroxyvitamin D and risk of post-menopausal breast cancer--results of a large case-control study. Carcinogenesis. 2008 Jan;29(1):93-9. doi: 10.1093/carcin/bgm240. Epub 2007 Oct 31. PMID 17974532
- [Result] Khan QJ, Reddy PS, Kimler BF, Sharma P, Baxa SE, O'Dea AP, Klemp JR, Fabian CJ. Effect of vitamin D supplementation on serum 25-hydroxy vitamin D levels, joint pain, and fatigue in women starting adjuvant letrozole treatment for breast cancer. Breast Cancer Res Treat. 2010 Jan;119(1):111-8. doi: 10.1007/s10549-009-0495-x. Epub 2009 Aug 5. PMID 19655244
- [Result] Peppone LJ, Huston AJ, Reid ME, Rosier RN, Zakharia Y, Trump DL, Mustian KM, Janelsins MC, Purnell JQ, Morrow GR. The effect of various vitamin D supplementation regimens in breast cancer patients. Breast Cancer Res Treat. 2011 May;127(1):171-7. doi: 10.1007/s10549-011-1415-4. Epub 2011 Mar 8. PMID 21384167
- [Result] Mann GB, Kang YC, Brand C, Ebeling PR, Miller JA. Secondary causes of low bone mass in patients with breast cancer: a need for greater vigilance. J Clin Oncol. 2009 Aug 1;27(22):3605-10. doi: 10.1200/JCO.2008.20.2549. Epub 2009 Jun 22. PMID 19546403
- [Derived] Chartron E, Firmin N, Touraine C, Chapelle A, Legouffe E, Rifai L, Pouderoux S, Roca L, D'Hondt V, Jacot W. A Phase II Multicenter Trial on High-Dose Vitamin D Supplementation for the Correction of Vitamin D Insufficiency in Patients with Breast Cancer Receiving Adjuvant Chemotherapy. Nutrients. 2021 Dec 10;13(12):4429. doi: 10.3390/nu13124429. PMID 34959982